CLINICAL TRIAL: NCT04557553
Title: Effects of Lagenbone on Improvements in Bone Mineral Density - A Pilot Study
Brief Title: Effects of Lagenbone on Bone Mineral Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Collaborators: Sun Ten Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Professor, Research Director, Southern California University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUNT001
Record Dates: First submitted 2020-04-30; First posted 2020-09-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Osteoporosis
Keywords: chinese medicine; herbal medicine; osteoporosis; bone mineral density
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lagenbone (Experimental): Lagenbone 500mg capsules, 8 capsules by mouth every day for 12 months.
  Interventions: Dietary Supplement: Lagenbone

INTERVENTIONS:
Dietary Supplement: Lagenbone — Traditional Chinese medicine herbal formula
  Other Names: Gui Lu Er Xian Jiao

SUMMARY:
To study the effects of the herbal supplement Lagenbone on Bone Mineral Density

DETAILED DESCRIPTION:
To study the effects of the herbal supplement Lagenbone on Bone Mineral Density. Lagenbone is a supplement based on the Chinese Herbal formula Gui Lu Er Xian Jiao.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of osteoporosis
* Able to read and understand English
* Willing to receive routine DEXA scans and comply with supplement schedule

Exclusion Criteria:

* Pregnant, lactating, or having gestational diabetes
* Diagnosed with comorbid conditions that they are taking medication for e.g. Acid reflux, Hashimoto's/Grave's Disease, Endometriosis, prostate, breast, uterine cancer, kidney disease, fibroids, psychological disorders
* Use of any medication known to interfere with bone mineral density
* Are taking any new medications/supplements/treatments/therapeutic exercise within the last two months for osteoporosis or bone density
* Involved in health-related litigation, claims
* Missing baseline visits
* Vegan or vegetarian
* Diagnosed with Alzheimer's or demonstrating onset of dementia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Dual-energy x-ray absorptiometry (DXA)DEXA Scan | 15 months
  Dual-energy x-ray absorptiometry (DXA) or bone densitometry or Bone Density Scan

SECONDARY OUTCOMES:
Short Osteoporosis Quality of Life Questionnaire (ECOS16) | 15 months
  Short Osteoporosis Quality of Life Questionnaire
36-item Short form survey (SF36) | 15 months
  36-item Short form survey
Osteoporotic Quality of Life Questionnaire (OQLQ10) | 15 months
  Osteoporotic Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Prasad S Vinjamury, DACM, MPH, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: No